CLINICAL TRIAL: NCT02333643
Title: A Phase 2, Randomized, Vehicle-Controlled, Double-Blind, Study to Evaluate Efficacy and Safety of Topical Ionic Contra-viral Therapy (ICVT) Comprised of CLS003 in Cutaneous Warts
Brief Title: A Phase 2 Efficacy Study of CLS003 ICVT in Subjects With Cutaneous Warts.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS003-CO-PR-002
Record Dates: First submitted 2014-12-19; First posted 2015-01-07 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Cutaneous Warts
MeSH Terms: interventions — Furosemide; Digoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CLS003 (Experimental): Topical digoxin/furosemide
  Interventions: Drug: CLS003
- Digoxin topical formulation (Experimental)
  Interventions: Drug: Digoxin
- Furosemide topical formulation (Experimental)
  Interventions: Drug: Furosemide
- Vehicle topical formulation (Placebo Comparator)
  Interventions: Drug: Vehicle topical

INTERVENTIONS:
Drug: CLS003
  Arms: CLS003
Drug: Furosemide
  Arms: Furosemide topical formulation
Drug: Digoxin
  Arms: Digoxin topical formulation
Drug: Vehicle topical
  Arms: Vehicle topical formulation

SUMMARY:
A phase 2, randomized, vehicle-controlled, double-blind study to assess the efficacy, safety and pharmacodynamics (PD) of topically applied CLS003 in otherwise healthy patients with cutaneous warts.

ELIGIBILITY:
Inclusion Criteria:

* absence of evidence of any active or chronic disease;
* Free of clinical significant systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of Adverse Events;
* Have at least 2 (non-subungual) common warts or at least 2 plantar warts on non-genital, nonfacial skin

Exclusion Criteria:

* Any clinically significant abnormality that in the opinion of the investigator would interfere with the study objectives or compromise subject safety;
* For women: a positive pregnancy test and/or nursing at screening or women who plan to become pregnant or are breastfeeding;
* A positive test for drugs of abuse at screening;
* History of alcohol or illicit drug abuse (alcohol abuse defined as alcohol consumption > 28 units/week);
* Positive test results for Hepatitis B, Hepatitis C or HIV;
* Have used salicylic acid or any other over-the-counter wart-removing product in the treatment area within 30 days prior to starting the study or cryotherapy within 60 days of starting the study;
* Have required systemic intake of immunosuppressive or immunomodulatory medication (including oral or parenteral corticosteroids) within 30 days prior to enrollment or during the course of the study. Routine use of inhaled or intranasal corticosteroids during the study is allowed;
* Have a known sensitivity to any of the investigational product ingredients
* Clinically relevant abnormal laboratory results, ECG, vital signs, or physical findings at screening;
* Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times in the past year;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in morphological wart assessment | Days 14, 28, 42, 70, 98
Change from baseline in Wart size and morphology assessment by standardized clinical photography | Days 14, 28, 42, 70, 98
Change from baseline in HPV viral load assessment of target lesions by quantitative PCR | Days 14, 28, 42, 70, 98
Reduction in wart size | Days 14, 28, 42, 70, 98
Change in the HPV viral load | Days 14, 28, 42, 70, 98
Change from baseline in mean HPV viral load | Days 14, 28, 42, 70, 98
Percent clearance of warts | Days 14, 28, 42, 70, 98

SECONDARY OUTCOMES:
Adverse event to evaluate safety and tolerability of CLS003 | Days 0-98

CONTACTS AND LOCATIONS:
Overall Officials: J. (Koos) Burggraaf, MD, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- LUMC/Centre for Human Drug Research, Leiden, Netherlands

REFERENCES:
- [Derived] Rijsbergen M, Niemeyer-van der Kolk T, Hogendoorn G, Kouwenhoven S, Lemoine C, Klaassen ES, de Koning M, Beck S, Bouwes Bavinck JN, Feiss G, Burggraaf J, Rissmann R. A randomized controlled proof-of-concept trial of digoxin and furosemide in adults with cutaneous warts. Br J Dermatol. 2019 May;180(5):1058-1068. doi: 10.1111/bjd.17583. Epub 2019 Mar 7. PMID 30580460